CLINICAL TRIAL: NCT01899469
Title: Efficiency of Physiotherapy Treatments for Low Back Pain in Women.
Acronym: LUMCRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Marta Romeu Ferran, SD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUMCRO
Record Dates: First submitted 2013-07-04; First posted 2013-07-15 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Magnetic Field Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Electromagnetic therapy (EM) (Experimental): The group had performed 20 sessions of EM therapy for 20 minutes and after had a 25 minutes from Back School intervention.
  Interventions: Procedure: Electromagnetic Therapy; Procedure: Back School
- Transcutaneous Electrical Neurological Stimulation (TENS) (Experimental): The group had performed 20 sessions of TENS therapy for 20 minutes and after had a 25 minutes from Back School intervention.
  Interventions: Procedure: Transcutaneous Electrical Neurological Stimulation; Procedure: Back School
- Back School (BS) (Experimental): The group had performed 20 sessions of Back School therapy for 25 minutes.
  Interventions: Procedure: Back School

INTERVENTIONS:
Procedure: Electromagnetic Therapy — 20 sessions from Monday to Friday of 20 minutes of Electromagnetic Therapy, using the next parameters: 10 Hz of frequency and 60% of intensity, and 20 sessions from Monday to Friday of 25 minutes of Back School, the exercises were based on the re-education of breathing, self stretching trunk muscles, erector spine reinforcement, abdominal reinforcement and postural exercises. The participants had been performing 8 to 10 repetitions of each exercise and they had been recommended about making a series more at home.
  Arms: Electromagnetic therapy (EM)
Procedure: Transcutaneous Electrical Neurological Stimulation — Procedure/Surgery: Transcutaneous Electrical Neurological Stimulation (TENS)
  20 sessions from Monday to Friday of 20 minutes of TENS Therapy using the next parameters: 100μs of impulse width, 80 Hz of impulse frequency, and 20 sessions from Monday to Friday of 25 minutes of Back School, the exercises were based on the re-education of breathing, self stretching trunk muscles, erector spine reinforcement, abdominal reinforcement and postural exercises. The participants had been performing 8 to 10 repetitions of each exercise and they had been recommended about making a series more at home.
  Arms: Transcutaneous Electrical Neurological Stimulation (TENS)
Procedure: Back School — 25 minutes of Back School, the exercises were based on the re-education of breathing, self stretching trunk muscles, erector spine reinforcement, abdominal reinforcement and postural exercises. The participants had been performing 8 to 10 repetitions of each exercise and they had been recommended about making a series more at home.

SUMMARY:
Aim: To evaluate and compare the effectiveness of a combined treatment of TENS or Elec-tromagnetic and Back School with the effectiveness of only the Back School treatment.

Design: Single-blind experimental prospective study of clinic intervention. Setting: Physiotherapy and Speech Therapy Unit at the Cambrils Slight Hospital. Spain.

Population: 96 women (50-85 years) with chronic low back pathology. Methods: Subjects were divided into three randomized groups: Back School (group 1), TENS with Back School (group 2), and Magnetic therapy with Back School (group 3). They have re-ceived 20 sessions of treatment. The intensity of pain (EVA Scale) and the quality of life (Oswestry Scale) were measured, at the beginning and at the end of the treatment and after three and six months. Anthropometric and physical activity variables were collected.

ELIGIBILITY:
Inclusion Criteria:

* Women between 50 and 85 years.
* Chronic LBP condition for at least three months ago.
* Patient's agreement by signing the consent.

Exclusion Criteria:

* Cardiac pacemaker carriers.
* Patients with parts of osteosynthesis and / or prostheses.
* Patients with a not well balanced medical condition.
* Patients with TENS at home and / or having completed physiotherapy during the last three months.
* Patients with skin infectious diseases or skin lesions and / or areas of hypoesthesia.
* Patients with malignant tumours.
* Patients who received any spinal injection during the last six weeks.
* Patients who participate or have participated in a study in the last three months

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain was measured at the beginning and after the treatment with the Visual Scale Analogue (VAS) | 24 weeks
  The VAS scale represents the pain intensity on a line of 10 cm, at one end there are the words "no pain" and the other end "the worst imaginable pain " written, the distance in centimetres from the "no pain" point to the place marked by the patient represents the intensity of pain
Oswestry disability index (ODI) | 24 weeks
  . The ODI assesses nine different aspects of disability, affecting various functions of daily life (personal care, lifting, walking, sitting, standing, sleeping, sex life, social life, and traveling). The questionnaire is scored using a global percentage score. For every section, one of six options is chosen. Each section is scored 0-5, with 0 indicating no limitation of function due to pain, and with 5 indicating major functional disability due to back pain.

SECONDARY OUTCOMES:
Questionnaire of Physical Activity (ClassAF) | 4 weeks
  Is a method developed by the Health Department of the Catalan Government. The ClassAf is a comprehensive questionnaire which contains a few items (1-4) to measure the general level of Physical Activity, it is calculated in METS (basal metabolic expenditure: mlO2/kg.min) and it allows to classify people into physically active or physically inactive.

OTHER OUTCOMES:
Body Mass Index (BMI) | 4 weeks
  On the basis of BMI (kg/m2), subjects were classified as Obesity (BMI over 30), overweight (BMI between 25 and 29.9) or normal weight (BMI between 18.5 and 24.9).

CONTACTS AND LOCATIONS:
Overall Officials: Ester Poblet, PT, Principal Investigator — University Rovira i Virgili
Locations (1):
- Hospital Lleuger de Cambrils, Cambrils, Tarragona, Spain